CLINICAL TRIAL: NCT00722605
Title: The Use of Multiple Respiration-Correlated Cone Beam CT Scans to Reduce Target Positioning Errors in Radiotherapy Treatment of Thoracic Cancer.
Brief Title: Multiple Respiration-Correlated Cone Beam Computed Tomography (CT) Scans to Reduce Target Positioning Errors in Radiotherapy Treatment of Thoracic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-080
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Esophageal Cancer; Lung Cancer
Keywords: lung; esophageal; cone beam ct scan
MeSH Terms: conditions — Esophageal Neoplasms; Lung Neoplasms

ARMS (1):
- 1 (Experimental): cone-beam CT based
  Interventions: Procedure: cone-beam CT

INTERVENTIONS:
Procedure: cone-beam CT — You will have the following CT scans along with the standard weekly portal images:Before treatment you will have a CT scan (a respiratory-correlated CT scan) at the time of the radiation planning, or simulation planning.During the first week of treatment - you will have 5 cone-beam CT scans at days 1 through 5 of your radiation treatment schedule.
  * During the remaining weeks of treatment - you will have a cone-beam CT scan every week. Depending on the number of treatments that your study doctor has prescribed for you, the number of weekly scans can be between 3 and 7.
  * For all scans, an external monitor will be used to record your breathing.
  * If needed, you will be repositioned by adjusting the radiation machine's treatment couch position.
  Other Names: The total number of cone-beam CT scans can be between 8 and 10. The scans will take about 15; minutes and will occur before your treatment. The scans will help determine whether the; radiation is being delivered accurately to the tumor and whether adjustments need to be made.

SUMMARY:
The purpose of this study is to use cone-beam CT scans to more accurately position the tumor during radiation and to see whether this method is more effective than the standard method of using 2D images (portal images), which is a type of X-ray. Cone-beam CT is a type of CT scanner attached to the treatment accelerator that produces 3D images of the patient.

The ability to eliminate the tumor with radiation depends in part on the accuracy of delivering the radiation to the lung. The position of the tumor changes because of normal breathing. Therefore, we want to improve the accuracy of the way the radiation is delivered to the tumor. With cone-beam CT scans taken before and during your treatment, we will be able to determine the location of the tumor with 3D images, measure how much the tumor moves as you breathe, and then position you so that the tumor will get the best delivery of radiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic proof of a thoracic malignancy, confirmed at MSKCC and suitable for radiation therapy, in order to be eligible for this study.
* Patients must be older than 18 years of age
* At least part of the tumor must be visible as observed in a diagnostic or planning CT. Patients must have Karnofsky Performance Status ≥ 70%

Exclusion Criteria:

* Pregnant Women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
To enhance the accuracy of treatment delivery by using a cone-beam CT guided patient positioning procedure, relative to the standard portal image guided procedure. | conclusion of the study

SECONDARY OUTCOMES:
To determine the reduction in the proportion of patients with large target positioning errors using the cone-beam CT guided procedure. | conclusion of the study
To gather data on organ motion and setup errors in the thorax and how they vary over the treatment course, in order to develop efficient clinical correction strategies. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Rimner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org